CLINICAL TRIAL: NCT07246785
Title: Efficacy of Anrikefon-based Patient-controlled Intravenous Analgesia for Pain Management After Laparoscopic Surgery: a Randomized, Double-blind, Active-controlled Pilot Trial
Brief Title: Anrikefon-based Patient-controlled Intravenous Analgesia After Laparoscopic Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anaesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025R0444
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Laparoscopic Surgery; Visceral Pain, Postoperative; Anrikefon; Patient-controlled Intravenous Analgesia
Keywords: Laparoscopic surgery; Visceral pain, Postoperative; Anrikefon; Patient-controlled intravenous analgesia
MeSH Terms: conditions — Visceral Pain | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High-dose anrikefon group (Experimental): Postoperative patient-controlled intravenous analgesia is established with anrikefon 1000 μg, diluted with normal saline to 100 ml, and programmed to administer an initial loading dose of 8 ml, followed by 4-ml boluses with a lockout interval of 10 minutes and no continuous background infusion.
  Interventions: Drug: High-dose anrikefon
- Medium-dose anrikefon group (Experimental): Postoperative patient-controlled intravenous analgesia is established with anrikefon 750 μg, diluted with normal saline to 100 ml, and programmed to administer an initial loading dose of 8 ml, followed by 4-ml boluses with a lockout interval of 10 minutes and no continuous background infusion.
  Interventions: Drug: Medium-dose anrikefon
- Low-dose anrikefon group (Experimental): Postoperative patient-controlled intravenous analgesia is established with anrikefon 500 μg, diluted with normal saline to 100 ml, and programmed to administer an initial loading dose of 8 ml, followed by 4-ml boluses with a lockout interval of 10 minutes and no continuous background infusion.
  Interventions: Drug: Low-dose anrikefon
- Morphine group (Active Comparator): Postoperative patient-controlled intravenous analgesia is established with morphine 50 mg, diluted with normal saline to 100 ml, and programmed to administer an initial loading dose of 8 ml, followed by 4-ml boluses with a lockout interval of 10 minutes and no continuous background infusion.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: High-dose anrikefon — Patients in this group receive postoperative patient-controlled intravenous analgesia for 48 hours. The formula comprises anrikefon (10 μg/ml), diluted with normal saline to 100 ml. The analgesic pump is set to deliver an initial loading dose of 8 ml, followed by patient-controlled boluses of 4 ml with a 10-minute lockout interval and no background infusion.
  Other Names: High-dose anrikefon-based patient-controlled analgesia
  Arms: High-dose anrikefon group
Drug: Medium-dose anrikefon — Patients in this group receive postoperative patient-controlled intravenous analgesia for 48 hours. The formula comprises anrikefon (7.5 μg/ml), diluted with normal saline to 100 ml. The analgesic pump is set to deliver an initial loading dose of 8 ml, followed by patient-controlled boluses of 4 ml with a 10-minute lockout interval and no background infusion.
  Other Names: Medium-dose anrikefon-based patient-controlled analgesia
  Arms: Medium-dose anrikefon group
Drug: Low-dose anrikefon — Patients in this group receive postoperative patient-controlled intravenous analgesia for 48 hours. The formula comprises anrikefon (5 μg/ml), diluted with normal saline to 100 ml. The analgesic pump is set to deliver an initial loading dose of 8 ml, followed by patient-controlled boluses of 4 ml with a 10-minute lockout interval and no background infusion.
  Other Names: Low-dose anrikefon-based patient-controlled analgesia
  Arms: Low-dose anrikefon group
Drug: Morphine — Patients in this group receive postoperative patient-controlled intravenous analgesia for 48 hours. The formula comprises morphine (0.5 mg/ml), diluted with normal saline to 100 ml. The analgesic pump is set to deliver an initial loading dose of 8 ml, followed by patient-controlled boluses of 4 ml with a 10-minute lockout interval and no background infusion.
  Other Names: Morphine-based patient-controlled analgesia
  Arms: Morphine group

SUMMARY:
Visceral pain following laparoscopic surgery is frequently underestimated, yet it is associated with a range of adverse outcomes. Effective visceral pain management should constitute an essential component of postoperative analgesic strategies following laparoscopic procedures. However, conventional analgesic agents, including μ-opioid receptor agonists, lack specificity for visceral pain. Anrikefon, a novel selective peripheral κ-opioid receptor agonist, demonstrates unique efficacy in alleviating visceral pain with a favorable safety profile. Preliminary studies showed that a single intravenous dose of anrikefon effectively alleviates postoperative pain after abdominal surgery with a low risk of adverse effects. The investigators hypothesize that an appropriate dosing regimen of anrikefon administered via patient-controlled intravenous analgesia (PCIA) pump, as part of a multimodal analgesic strategy, can specifically target and alleviate visceral pain after laparoscopic surgery, thereby achieving comprehensive postoperative analgesia.

DETAILED DESCRIPTION:
Approximately 50% to 90% of patients undergoing abdominal surgery experience moderate or severe acute postoperative pain, which primarily comprises somatic, visceral, and inflammatory pain components, with peak intensity typically occurring within the first 24 to 72 hours after surgery. Inadequate management of acute postoperative pain not only increases patients' suffering and impairs their sleep quality, but also increases the risk of postoperative complications, delays postsurgical recovery, prolongs hospital stay, elevates healthcare costs, and even contributes to the development of chronic neuropathic pain.

With advances in minimally invasive techniques and the widespread application of laparoscopic surgery, surgical incisions on the body surface have been significantly reduced, leading to diminished somatic pain. However, the intra-abdominal visceral injury is not necessarily reduced and can even be more substantial in this context, leading to prominent postoperative visceral pain that perioperative clinicians often underestimate. Consequently, effective management of visceral pain should be an essential component of postoperative analgesic strategies following laparoscopic procedures.

Opioids, renowned for their potent analgesic efficacy, serve as the cornerstone of perioperative acute pain management and constitute a critical element of multimodal analgesic regimens. Nevertheless, due to the sparse expression of μ-opioid receptors in visceral pain pathways and their weak modulation of visceral pain afferent signaling, the conventional μ-opioid receptor agonists, such as morphine, exhibit limited effectiveness against visceral pain. Anrikefon is a novel selective peripheral κ-opioid receptor agonist. Due to the high expression levels of κ-opioid receptors within visceral pain pathways, anrikefon exerts an unique therapeutic effect in alleviating visceral pain with a relatively low risk of adverse effects.

Preliminary studies indicate that a single intravenous dose of Anrikefon effectively alleviates pain after abdominal surgery with a low incidence of adverse effects. Additional evidence suggests that patient-controlled intravenous administration of anrikefon provides effective analgesia after orthopedic surgery without respiratory depression or other severe adverse effects. However, the appropriate dosing regimen of anrikefon for patient-controlled intravenous analgesia (PCIA) following laparoscopic surgery remains to be established.

The investigators hypothesize that administering appropriate doses of anrikefon via PCIA pump, as part of a multimodal analgesic regimen that comprises regional nerve blocks targeting somatic pain and nonsteroidal anti-inflammatory drugs (NSAIDs) targeting inflammatory pain, will specifically and effectively alleviate visceral pain following laparoscopic surgery. This pilot trial aims to explore the preliminary efficacy and optimal dosing regimen of anrikefon administered via PCIA after laparoscopic surgery, assess the feasibility of conducting a larger-scale randomized controlled trial, and provide essential parameters for sample size estimation in subsequent investigations.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years but < 75 years;
2. Scheduled to undergo elective laparoscopic gastrointestinal surgery with an expected duration of ≥1 hour;
3. The incisional pain can be covered by the transversus abdominis plane block or rectus sheath block; yet patients still require postoperative patient-controlled intravenous analgesia.

Exclusion Criteria:

1. Presence of preoperative cognitive impairment (Mini-Mental State Examination [MMSE] score < 27), or inability to communicate due to language barrier;
2. Body mass index (BMI) > 30 kg/m² or < 18 kg/m²;
3. Presence of poorly controlled or untreated comorbidities, including but not limited to the following: hypertension characterized by a resting systolic blood pressure (SBP) > 180 mmHg and/or diastolic blood pressure (DBP) > 110 mmHg, coronary artery disease with unstable angina or myocardial infarction within 6 months, heart failure rated as New York Heart Association classification ≥ III, severe chronic obstructive pulmonary disease (or in a state of acute exacerbation), severe hepatic insufficiency (Child-Pugh grade C), severe renal insufficiency (estimated glomerular filtration rate < 30 ml/min/1.73m²), or American Society of Anesthesiologists (ASA) physical status classification ≥ IV;
4. Continuous use of opioid analgesics for more than 10 days for any reason, or alcohol abuse (average daily intake of pure alcohol > 36 g) within 3 months before screening;
5. Preoperative use of opioid or non-opioid analgesics with the interval between the last administration and randomization shorter than five half-lives of the drug or the duration of drug action (whichever is longer);
6. Known allergies or contraindications to opiates or other medications that may be used in this study, such as anesthetics, antiemetics, and nonsteroidal anti-inflammatory drugs (NSAIDs);
7. Anticipated need for postoperative mechanical ventilation；
8. Other conditions that are considered unsuitable for study participation.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-12-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Time-weighted sum of pain intensity difference (SPID) of movement-evoked visceral pain within 48 hours | Within 48 hours after intervention.
  Time-weighted SPID is defined as the cumulative sum of the product obtained by multiplying the pain intensity difference at each time point (calculated by subtracting the baseline pain intensity score from the current pain intensity score) by the time difference (the current time point minus the previous time point). Movement-evoked visceral pain intensity will be assessed before intervention and at 0.5, 1, 2, 6, 12, 24, 36, and 48 hours after intervention using an 11-point Numeric Rating Scale (0 = no pain, 10 = the worst pain).

SECONDARY OUTCOMES:
Time-weighted SPID of visceral pain at rest within 48 hours | Within 48 hours after intervention.
  Time-weighted SPID is defined as the cumulative sum of the product obtained by multiplying the pain intensity difference at each time point (calculated by subtracting the baseline pain intensity score from the current pain intensity score) by the time difference (the current time point minus the previous time point). The intensity of visceral pain at rest will be assessed before intervention and at 0.5, 1, 2, 6, 12, 24, 36, and 48 hours after intervention using an 11-point Numeric Rating Scale (0 = no pain, 10 = the worst pain).
Time-weighted SPID of movement-evoked somatic pain within 48 hours | Within 48 hours after intervention.
  Time-weighted SPID is defined as the cumulative sum of the product obtained by multiplying the pain intensity difference at each time point (calculated by subtracting the baseline pain intensity score from the current pain intensity score) by the time difference (the current time point minus the previous time point). Movement-evoked somatic pain intensity will be assessed before intervention and at 0.5, 1, 2, 6, 12, 24, 36, and 48 hours after intervention using an 11-point Numeric Rating Scale (0 = no pain, 10 = the worst pain).
Time-weighted SPID of somatic pain at rest within 48 hours | Within 48 hours after intervention.
  Time-weighted SPID is defined as the cumulative sum of the product obtained by multiplying the pain intensity difference at each time point (calculated by subtracting the baseline pain intensity score from the current pain intensity score) by the time difference (the current time point minus the previous time point). The intensity of somatic pain at rest will be assessed before intervention and at 0.5, 1, 2, 6, 12, 24, 36, and 48 hours after intervention using an 11-point Numeric Rating Scale (0 = no pain, 10 = the worst pain).
Time-weighted SPID of movement-evoked overall pain within 48 hours | Within 48 hours after intervention.
  Time-weighted SPID is defined as the cumulative sum of the product obtained by multiplying the pain intensity difference at each time point (calculated by subtracting the baseline pain intensity score from the current pain intensity score) by the time difference (the current time point minus the previous time point). Movement-evoked overall pain intensity will be assessed before intervention and at 0.5, 1, 2, 6, 12, 24, 36, and 48 hours after intervention using an 11-point Numeric Rating Scale (0 = no pain, 10 = the worst pain).
Time-weighted SPID of overall pain at rest within 48 hours | Within 48 hours after intervention.
  Time-weighted SPID is defined as the cumulative sum of the product obtained by multiplying the pain intensity difference at each time point (calculated by subtracting the baseline pain intensity score from the current pain intensity score) by the time difference (the current time point minus the previous time point). The intensity of overall pain at rest will be assessed before intervention and at 0.5, 1, 2, 6, 12, 24, 36, and 48 hours after intervention using an 11-point Numeric Rating Scale (0 = no pain, 10 = the worst pain).

OTHER OUTCOMES:
Quality of recovery at 24 hours after surgery | At the 24th hour after surgery.
  Quality of postoperative recovery is assessed using the 15-item Quality of Recovery (QoR-15) scale, a patient-reported questionnaire that evaluates recovery after anesthesia and surgery across five domains: physical comfort, emotional state, psychological support, pain, and activities of daily living. The total score ranges from 0 to 150, with higher scores indicating better quality of postoperative recovery.
Number of patient-controlled analgesia (PCA) attempts within 48 hours after intervention | Within 48 hours after intervention.
  The total count of times a patient presses the PCA button to self-administer analgesics.
Rate of rescue analgesia within 48 hours after intervention | Within 48 hours after intervention.
  The proportion of patients who require supplemental analgesics.
Patient satisfaction with postoperative analgesia at 48 hours after intervention | At the 48th hour after intervention.
  Patient satisfaction with postoperative analgesia will be evaluated at the 48th hour after intervention, using an 11-point Numeric Rating Scale (0 = the lowest level of satisfaction, 10 = the highest level of satisfaction).
Subjective sleep quality on the night of surgery and the first postoperative night | From the night of surgery until the first night after surgery.
  Subjective sleep quality during the previous night will be assessed the next morning (between 8:00 and 10:00 am) using an 11-point Numeric Rating Scale (0 = the best sleep, 10 = the worst sleep).
Time to first flatus and time to first defecation | Up to 30 days after surgery.
  Time to first flatus and time to first defecation.
Time to first ambulation | Up to 30 days after surgery.
  Time to first walking on the ground after surgery.
Length of stay in hospital after surgery | Up to 30 days after surgery.
  Length of stay in hospital after surgery.
Incidence of postoperative complications (including all-cause mortality) within 30 days after surgery | Up to 30 days after surgery.
  Postoperative complications are defined as new-onset medical events that are harmful to patients' recovery and require therapeutic interventions, that is grade II or higher based on the Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu Y, Xiao S, Yang H, Lv X, Hou A, Ma Y, Jiang Y, Duan C, Mi W; CAPOPS Group. Postoperative pain-related outcomes and perioperative pain management in China: a population-based study. Lancet Reg Health West Pac. 2023 Jun 10;39:100822. doi: 10.1016/j.lanwpc.2023.100822. eCollection 2023 Oct. PMID 37927993
- [Background] Armstrong RA, Fayaz A, Manning GLP, Moonesinghe SR; Peri-operative Quality Improvement Programme (PQIP) delivery team; Oliver CM; PQIP collaborative. Predicting severe pain after major surgery: a secondary analysis of the Peri-operative Quality Improvement Programme (PQIP) dataset. Anaesthesia. 2023 Jul;78(7):840-852. doi: 10.1111/anae.15984. Epub 2023 Mar 2. PMID 36862937
- [Background] Glare P, Aubrey KR, Myles PS. Transition from acute to chronic pain after surgery. Lancet. 2019 Apr 13;393(10180):1537-1546. doi: 10.1016/S0140-6736(19)30352-6. PMID 30983589
- [Background] Wildbrett P, Oh A, Naundorf D, Volk T, Jacobi CA. Impact of laparoscopic gases on peritoneal microenvironment and essential parameters of cell function. Surg Endosc. 2003 Jan;17(1):78-82. doi: 10.1007/s00464-002-9015-3. Epub 2002 Sep 30. PMID 12360379
- [Background] Papparella A, Noviello C, Romano M, Parmeggiani P, Paciello O, Papparella S. Local and systemic impact of pneumoperitoneum on prepuberal rats. Pediatr Surg Int. 2007 May;23(5):453-7. doi: 10.1007/s00383-006-1860-z. PMID 17333216
- [Background] Hatipoglu S, Akbulut S, Hatipoglu F, Abdullayev R. Effect of laparoscopic abdominal surgery on splanchnic circulation: historical developments. World J Gastroenterol. 2014 Dec 28;20(48):18165-76. doi: 10.3748/wjg.v20.i48.18165. PMID 25561784
- [Background] de Lacy FB, Taura P, Arroyave MC, Trepanier JS, Rios J, Bravo R, Ibarzabal A, Pena R, Deulofeu R, Lacy AM. Impact of pneumoperitoneum on intra-abdominal microcirculation blood flow: an experimental randomized controlled study of two insufflator models during transanal total mesorectal excision : An experimental randomized multi-arm trial with parallel treatment design. Surg Endosc. 2020 Oct;34(10):4494-4503. doi: 10.1007/s00464-019-07236-5. Epub 2019 Nov 7. PMID 31701284
- [Background] Cheong JY, Keshava A, Witting P, Young CJ. Effects of Intraoperative Insufflation With Warmed, Humidified CO2 during Abdominal Surgery: A Review. Ann Coloproctol. 2018 Jun;34(3):125-137. doi: 10.3393/ac.2017.09.26. Epub 2018 Jun 30. PMID 29991201
- [Background] Sikandar S, Dickenson AH. Visceral pain: the ins and outs, the ups and downs. Curr Opin Support Palliat Care. 2012 Mar;6(1):17-26. doi: 10.1097/SPC.0b013e32834f6ec9. PMID 22246042
- [Background] Kendall GP. Visceral pain. Br J Surg. 1985 Sep;72 Suppl:S4-5. doi: 10.1002/bjs.1800721304. No abstract available. PMID 3899257
- [Background] Golzari SE, Nader ND, Mahmoodpoor A. Underlying Mechanisms of Postoperative Pain After Laparoscopic Surgery. JAMA Surg. 2016 Mar;151(3):295-6. doi: 10.1001/jamasurg.2015.3934. No abstract available. PMID 26535957
- [Background] Choi JB, Kang K, Song MK, Seok S, Kim YH, Kim JE. Pain Characteristics after Total Laparoscopic Hysterectomy. Int J Med Sci. 2016 Jul 5;13(8):562-8. doi: 10.7150/ijms.15875. eCollection 2016. PMID 27499688
- [Background] Blichfeldt-Eckhardt MR, Ording H, Andersen C, Licht PB, Toft P. Early visceral pain predicts chronic pain after laparoscopic cholecystectomy. Pain. 2014 Nov;155(11):2400-7. doi: 10.1016/j.pain.2014.09.019. Epub 2014 Sep 22. PMID 25250720
- [Background] Ruiz-Tovar J, Garcia A, Ferrigni C, Duran M. Application of Vitamin E Acetate on Staple Lines and Anastomoses of Roux-en-Y Gastric Bypass: Impact on Postoperative Pain and Acute Phase Reactants. Obes Surg. 2020 Aug;30(8):2988-2993. doi: 10.1007/s11695-020-04635-9. PMID 32342266
- [Background] Koh JC, Kong HJ, Kim MH, Hong JH, Seong H, Kim NY, Bai SJ. Comparison of Analgesic and Adverse Effects of Oxycodone- and Fentanyl-Based Patient-Controlled Analgesia in Patients Undergoing Robot-Assisted Laparoscopic Gastrectomy Using a 55:1 Potency Ratio of Oxycodone to Fentanyl: A Retrospective Study. J Pain Res. 2020 Sep 4;13:2197-2204. doi: 10.2147/JPR.S264764. eCollection 2020. PMID 32943912
- [Background] Jiang Z, Zhou G, Song Q, Bao C, Wang H, Chen Z. Effect of Intravenous Oxycodone in Combination With Different Doses of Dexmedetomdine on Sleep Quality and Visceral Pain in Patients After Abdominal Surgery: A Randomized Study. Clin J Pain. 2018 Dec;34(12):1126-1132. doi: 10.1097/AJP.0000000000000645. PMID 30134283
- [Background] Ehrlich AT, Kieffer BL, Darcq E. Current strategies toward safer mu opioid receptor drugs for pain management. Expert Opin Ther Targets. 2019 Apr;23(4):315-326. doi: 10.1080/14728222.2019.1586882. Epub 2019 Mar 15. PMID 30802415
- [Background] Waldhoer M, Bartlett SE, Whistler JL. Opioid receptors. Annu Rev Biochem. 2004;73:953-90. doi: 10.1146/annurev.biochem.73.011303.073940. PMID 15189164
- [Background] Beck TC, Hapstack MA, Beck KR, Dix TA. Therapeutic Potential of Kappa Opioid Agonists. Pharmaceuticals (Basel). 2019 Jun 20;12(2):95. doi: 10.3390/ph12020095. PMID 31226764
- [Background] Wang X, Gou X, Yu X, Bai D, Tan B, Cao P, Qian M, Zheng X, Wang H, Tang P, Zhang C, Ye F, Ni J. Antinociceptive and Antipruritic Effects of HSK21542, a Peripherally-Restricted Kappa Opioid Receptor Agonist, in Animal Models of Pain and Itch. Front Pharmacol. 2021 Nov 16;12:773204. doi: 10.3389/fphar.2021.773204. eCollection 2021. PMID 34867403
- [Background] Zhong Y, Xu Y, Lei Q, Yang M, Wang S, Hu X, Xie H, Li Y, Qin Z, Gu Z, Zhang J, Wang Y, Wu J, Wang H, Ming Y, Xia Z, Zhai H, Jiang K, Zhang P, Wang Z, Wang L, Li L, Cheng Z, Jiang H, Wang G, Chen J, Zhao Z, Chen X, Yan M. HSK21542 in patients with postoperative pain: two phase 3, multicentre, double-blind, randomized, controlled trials. Nat Commun. 2025 May 24;16(1):4830. doi: 10.1038/s41467-025-60013-y. PMID 40413233
- [Background] Shao R, Wang HY, Ruan ZR, Jiang B, Yang DD, Hu Y, Xu YC, Yang JT, Gao W, Zhao WY, Yan M, Lou H. Phase I clinical trial evaluating the safety, tolerance, pharmacokinetics and pharmacodynamics of HSK21542 injection in healthy volunteers. Basic Clin Pharmacol Toxicol. 2024 Dec;135(6):743-754. doi: 10.1111/bcpt.14094. Epub 2024 Oct 13. PMID 39397291
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542